CLINICAL TRIAL: NCT03217890
Title: Distribution Of ABO Blood Groups In Relation To Cleft Lip And/or Palate .
Brief Title: the Relationship Between Cleft Lip and / or Palate (Different Types) and ABO Blood Groups.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa medhat helmy, postgraduated student, Cairo University
Other Study IDs: CEBC-CU-2017-07-18
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Direct benefit of the research to assess the relationship between cleft lip and / or palate (different types) and ABO blood groups.

DETAILED DESCRIPTION:
376 Egyptian cleft lip and/or palate patients ( age ranged from 2 days to 15 years ) With no syndrome. Blood group from records will be collected an d then assess the relationship between cleft lip and / or palate (different types) and ABO blood groups.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian Patients with cleft or/and palate
* The children's age ranged between 2 days and 15 years.

Exclusion Criteria:

* syndromic patients

Ages: 2 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 376 Egyptian cleft lip and/or palate patients (Age ranged from 2 days to 15 years ) With no syndrome .
Sampling Method: Probability Sample
Enrollment: 376 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Distribution of ABO blood group in relation to different types of cleft lip and/or palate . | 6 months
  ABO blood group

IPD SHARING:
Plan to Share IPD: Undecided